CLINICAL TRIAL: NCT06813586
Title: DataNetCP: Establishing a Hospital-based Cerebral Palsy Registry in Italy
Brief Title: Observational Study for the Epidemiology of Cerebral Palsy in Italy
Acronym: DataNetCP
Status: Recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Fondazione Pierfranco e Luisa Mariani (Unknown); Fondazione FightTheStroke (Unknown); Istituto Superiore di Sanità (Other); IRCCS Eugenio Medea (Other); Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Principal Investigator, Giuseppina Sgandurra, Associate Professor, Head of INNOVATE Lab, IRCCS Fondazione Stella Maris
Other Study IDs: DataNetCP
Record Dates: First submitted 2025-01-28; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Database; Hospital-based registry
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with CP: Children with diagnosed CP age: 4-18 years old
  Interventions: Other: hospital-based registry

INTERVENTIONS:
Other: hospital-based registry — The clinical data collected for each patient will reflect comprehensive multiprofessional clinical insights necessary for diagnostic definition and typically obtained during diagnostic evaluation and/or monitoring visits. In addition to these, instrumental data commonly acquired in clinical practice, such as neuroradiological and electrophysiological information, will also be collected.
  For each enrolled subject, a checklist (CRF) will be completed to gather study-related data. These data will be entered into a specific database constructed on the REDCap platform and managed in an anonymized form. Subject enrollment will be conducted progressively.
  This data collection will enable monitoring of study progress, including the number of enrolled subjects, completed assessments, and study adherence. Every three months, monitoring will be performed to assess study progress and the achievement of enrollment targets.

SUMMARY:
BACKGROUND AND RATIONALE Cerebral Palsy (CP) is the leading cause of childhood disability, with an estimated prevalence of 2 to 2.5 per 1,000 births. This complex clinical condition encompasses motor development disorders as well as sensory, communication, cognitive, and emotional impairments. Despite the significant healthcare impact of CP, standardized guidelines for its study and treatment are lacking both nationally and internationally. Existing literature is limited by small sample sizes, inconsistent assessment tools, and insufficient etiopathogenetic and functional characterizations of different CP types. A national registry, which could offer comprehensive epidemiological data, does not currently exist.

This project aims to create a shared digital platform across clinical centers throughout Italy (three coordinative centers for northern, central, and southern Italy). This platform will allow systematic, standardized, retrospective, and prospective data collection, including clinical, instrumental, and genetic data (where available) for patients with CP. The study intends to complement ongoing national projects, such as the "Italian Network for Early Detection and Intervention in Developmental Disabilities (INEED)" and the "Italian Network for Cerebral Palsy (Ita-Net-CP)."

STUDY OBJECTIVES

This study aims to analyze epidemiological data, specifically:

* Evaluating the prevalence of various clinical types of CP
* Assessing the distribution of functional impairment severity and associated comorbidities.

STUDY DESIGN This is a non-profit, multicenter, observational study involving a cohort of CP patients, promoted within the Mariani Foundation Network. The study involves both retrospective and prospective data collection. It will enroll both patients already under care for follow-up and newly diagnosed patients.

A sample of at least 300 children and/or adolescents with CP of various etiologies, with 100 participants per clinical center, is targeted. Enrollment will be voluntary, either by invitation from the referring physician, who will explain the importance of the registry, or through project dissemination, allowing parents to request their children's inclusion. Basic registry items can be filled out by parents and, with permission, the primary physician for clinical fields. Parents can opt to be included in the registry to receive information on national clinical studies, approved by ethics committees.

Collected essential data includes:

* Identification and contact information for patient pseudonymization
* Socioeconomic status
* CP classification according to the European Surveillance Group
* Anamnesis regarding disorder etiology
* Neuroradiological classification based on SCPE (MRICS)
* Functional impairment level of each child
* Significant comorbidities

STUDY POPULATION At least 300 pediatric CP patients aged 4-18 years are expected to be recruited. Exclusion criteria only include lack of informed consent.

DRUG, MEDICAL DEVICE, NUTRACEUTICAL, BIOLOGICAL SAMPLES, OTHER ELEMENTS This observational study involves systematic, standardized retrospective and prospective data collection of clinical, instrumental, and genetic data (if available). No medical devices, pharmaceuticals, or nutraceuticals will be used. No human biological samples will be collected.

STUDY TIMELINE Study duration per patient: aligned with routine clinical visits. No additional evaluations are foreseen.

Recruitment duration: 12 months Overall study duration: 36 months

SAMPLE SIZE AND DATA ANALYSIS The study aims to recruit at least 300 pediatric CP patients. A control group is not planned.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy (CP) confirmed clinically in accordance with recent international guidelines (SCPE Guidelines, 2019);
* Age between 4 and 18 years.

Exclusion Criteria:

* Progressive neuromotor disorder (defined as a condition involving the loss of previously acquired abilities);
* Patients with a neurological condition defined by isolated hypotonia;
* Patients with neurological deficits secondary to spinal injury;

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population is expected to include at least 300 pediatric patients with cerebral palsy (CP) in accordance with the inclusion and exclusion criteria outlined by the SCPE Collaborative Group (2000).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Participants demographic data | Baseline
  Age, gender, birth date, place of birth, nationality, address (country)
Cerebral palsy (CP) classification | Baseline
  Classification of CP according to the European Surveillance Group (SCPE Guidelines, 2019):
  Spastic CP (bilateral or unilateral forms); Dyskinetic CP (dystonic form or choreoathetotic form); Ataxic CP.
Anamnestic data related to the etiopathogenesis of the disorder | Baseline
  This refers to the medical history and background information that help in understanding the cause and development of a disorder i.e. visual and auditory impairments, birth weight, cognitive level, epilepsy, Apgar score and comorbidities.
Level of Gross Motor Function Classification System (GMFCS) | Baseline
  The Gross Motor Function Classification System (GMFCS), is a five-level classification that differentiates children with cerebral palsy based on the child's current gross motor abilities, limitations in gross motor function, and need for assistive technology and wheeled mobility (Rosenbaum et al., 2008).
Level of Manual Ability Classification System (MACS) | Baseline
  Manual Ability Classification System (MACS) classifies the child's ability from 4 to 18 years old to handle objects in daily activities on one of 5 levels (level I: greater ability, level V: less ability). MACS level I (able to handle objects easily and successfully), level II (able to handle most objects but with somewhat reduced quality and/or speed of achievement so that alternate ways of performance might be used), level III (handles objects with difficulty; needs help to prepare and/or modify activities), level IV (needs continuous support, handles a limited selection of objects), level V (does not handle objects, needs total assistance) (Eliasson et al., 2006).
Level of Bimanual Fine Motor Function (BFMF) | Baseline
  Bimanual Fine Motor Function (BFMF) classifies fine motor function according to the child's best ability (capacity) to grasp, hold and manipulate objects for each hand separately. BFMF can be used in children from 3-18 years of age (Elvrum et al., 2016).
Level of Visual Function Classification System (VFCS) | Baseline
  The Visual Function Classification System (VFCS) is a tool used to classify the level of visual function in individuals with disabilities, particularly in the context of cerebral palsy. It is divided into five levels, each describing the degree of visual ability and the impact on daily activities (Baranello et al., 2020).
Level of Communication Function Classification System (CFCS) | Baseline
  The Communication Function Classification System (CFCS) is a classification tool used to assess and categorize the communication abilities of individuals with cerebral palsy or similar disabilities. It is divided into five levels, each describing the individual's ability to communicate in different environments with both familiar and unfamiliar partners.
Level of Viking Speech Scale (VSS) | Baseline
  The Viking Speech Scale (VSS) is a classification system designed to assess and categorize the speech abilities of individuals with cerebral palsy or other neurological conditions that affect communication. It focuses on the clarity and intelligibility of speech, as well as the individual's ability to communicate effectively with others. The scale is divided into four levels (Pennington et al., 2013).
Level of Eating and Drinking Classification System (EDACS) | Baseline
  The Eating and Drinking Classification System (EDACS) is a tool used to classify the eating and drinking abilities of individuals with disabilities, particularly in the context of cerebral palsy. It categorizes individuals into different levels based on their ability to safely and efficiently eat and drink, with a focus on both the safety and efficiency of these activities. The system is divided into five levels (Sellers et al., 2014).
Neuroradiological classification according to the classification promoted by SCPE (MRICS) | Baseline
  Magnetic Resonance Imaging Classification System is used in the context of neuroradiological assessment in cerebral palsy.
  A. Maldevelopments A.1. Disorders of cortical formation (proliferation and/or migration and/or organization A.2. Other maldevelopments (examples: holoprosencephaly Dandy-Walker malformation, corpus callosum agenesis, cerebellar hypoplasia) B. Predominant white matter injury B.1. PVL (mild/severe) B.2. Sequelae of IVH or periventricular haemorrhagic infarction B.3. Combination of PVL and IVH sequelae C. Predominant grey matter injury C.1. Basal ganglia/thalamus lesions (mild/moderate/severe) C.2. Cortico-subcortical lesions only (watershed lesions in parasagittal distribution/multicystic encephalomalacia) not covered under C3 C.3. Arterial infarctions (middle cerebral artery/other) D. Miscellaneous (examples: cerebellar atrophy, cerebral atrophy, delayed myelination, ventriculomegaly not covered under B, haemorrhage not covered under B, brainstem lesions, calcific

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Associazione La Nostra Famiglia - IRCCS Eugenio Medea, Brindisi, Apulia
  - Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan, Lombardy
  - IRCCS Fondazione Stella Maris, Calambrone, Tuscany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pennington L, Virella D, Mjoen T, da Graca Andrada M, Murray J, Colver A, Himmelmann K, Rackauskaite G, Greitane A, Prasauskiene A, Andersen G, de la Cruz J. Development of The Viking Speech Scale to classify the speech of children with cerebral palsy. Res Dev Disabil. 2013 Oct;34(10):3202-10. doi: 10.1016/j.ridd.2013.06.035. Epub 2013 Jul 24. PMID 23891732
- [Background] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461
- [Background] Baranello G, Signorini S, Tinelli F, Guzzetta A, Pagliano E, Rossi A, Foscan M, Tramacere I, Romeo DMM, Ricci D; VFCS Study Group. Visual Function Classification System for children with cerebral palsy: development and validation. Dev Med Child Neurol. 2020 Jan;62(1):104-110. doi: 10.1111/dmcn.14270. Epub 2019 Jun 10. PMID 31180136
- [Background] Himmelmann K, Horber V, De La Cruz J, Horridge K, Mejaski-Bosnjak V, Hollody K, Krageloh-Mann I; SCPE Working Group. MRI classification system (MRICS) for children with cerebral palsy: development, reliability, and recommendations. Dev Med Child Neurol. 2017 Jan;59(1):57-64. doi: 10.1111/dmcn.13166. Epub 2016 Jun 21. PMID 27325153
- [Background] Sellers D, Mandy A, Pennington L, Hankins M, Morris C. Development and reliability of a system to classify the eating and drinking ability of people with cerebral palsy. Dev Med Child Neurol. 2014 Mar;56(3):245-51. doi: 10.1111/dmcn.12352. Epub 2013 Dec 18. PMID 24344767
- [Background] Fiori S, Cioni G, Klingels K, Ortibus E, Van Gestel L, Rose S, Boyd RN, Feys H, Guzzetta A. Reliability of a novel, semi-quantitative scale for classification of structural brain magnetic resonance imaging in children with cerebral palsy. Dev Med Child Neurol. 2014 Sep;56(9):839-45. doi: 10.1111/dmcn.12457. Epub 2014 Apr 19. PMID 24750109
- [Background] Elvrum AK, Andersen GL, Himmelmann K, Beckung E, Ohrvall AM, Lydersen S, Vik T. Bimanual Fine Motor Function (BFMF) Classification in Children with Cerebral Palsy: Aspects of Construct and Content Validity. Phys Occup Ther Pediatr. 2016;36(1):1-16. doi: 10.3109/01942638.2014.975314. Epub 2014 Nov 6. PMID 25374154
- [Background] Eliasson AC, Krumlinde-Sundholm L, Rosblad B, Beckung E, Arner M, Ohrvall AM, Rosenbaum P. The Manual Ability Classification System (MACS) for children with cerebral palsy: scale development and evidence of validity and reliability. Dev Med Child Neurol. 2006 Jul;48(7):549-54. doi: 10.1017/S0012162206001162. PMID 16780622
- [Background] Long HL, Mahr TJ, Natzke P, Rathouz PJ, Hustad KC. Longitudinal change in speech classification between 4 and 10 years in children with cerebral palsy. Dev Med Child Neurol. 2022 Sep;64(9):1096-1105. doi: 10.1111/dmcn.15198. Epub 2022 Mar 9. PMID 35262181
- [Background] Rosenbaum PL, Palisano RJ, Bartlett DJ, Galuppi BE, Russell DJ. Development of the Gross Motor Function Classification System for cerebral palsy. Dev Med Child Neurol. 2008 Apr;50(4):249-53. doi: 10.1111/j.1469-8749.2008.02045.x. Epub 2008 Mar 1. PMID 18318732
- [Background] Sellier E, Surman G, Himmelmann K, Andersen G, Colver A, Krageloh-Mann I, De-la-Cruz J, Cans C. Trends in prevalence of cerebral palsy in children born with a birthweight of 2,500 g or over in Europe from 1980 to 1998. Eur J Epidemiol. 2010 Sep;25(9):635-42. doi: 10.1007/s10654-010-9474-0. Epub 2010 Jun 8. PMID 20532622
- [Background] Scheck SM, Pannek K, Fiori S, Boyd RN, Rose SE. Quantitative comparison of cortical and deep grey matter in pathological subtypes of unilateral cerebral palsy. Dev Med Child Neurol. 2014 Oct;56(10):968-75. doi: 10.1111/dmcn.12461. Epub 2014 Apr 19. PMID 24749496
- [Background] Surveillance of Cerebral Palsy in Europe. Surveillance of cerebral palsy in Europe: a collaboration of cerebral palsy surveys and registers. Surveillance of Cerebral Palsy in Europe (SCPE). Dev Med Child Neurol. 2000 Dec;42(12):816-24. doi: 10.1017/s0012162200001511. PMID 11132255